CLINICAL TRIAL: NCT05070871
Title: A Randomized, Double-blind Clinical Trial Investigating the Effect of Salmon Bone Meal on Osteoarthritis Among Men and Women
Brief Title: A Clinical Trial Investigating the Effect of Salmon Bone Meal on Osteoarthritis Among Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hofseth Biocare ASA (Industry)
Collaborators: Møre og Romsdal Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CALGO-ART
Record Dates: First submitted 2021-09-23; First posted 2021-10-07 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: stiffness; pain; knee pain; hip pain; osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrolyzed Collagen type II (Active Comparator): 10 capsules daily of hydrolyzed collagen (CH) type II is taken per orally. Each capsule contains ~500 mg of CH. Once or twice daily dosing. Duration: 6 months.
  Interventions: Dietary Supplement: Hydrolyzed Collagen
- Maltodextrin (Placebo Comparator): 10 capsules daily of maltodextrin is taken per orally. Each capsule contains 500 mg of maltodextrin. Once or twice daily dosing. Duration: 6 months.
  Interventions: Other: Placebo
- Unhydrolyzed Collagen type II (Salmon bone meal) (Experimental): 10 capsules daily of salmon bone meal enriched with vitamin D3 is taken per orally. Each capsule contains 300 mg of maltodextrin, 200 mg of salmon bone meal (10 capsules = 2000 mg salmon bone meal = 340 mg elemental calcium in the form of microcrystalline hydroxyapatite), and 4 micrograms of vitamin D3 (10 capsules = 40 micrograms of vitamin D3 = 1600 IU).
  Interventions: Dietary Supplement: CalGo

INTERVENTIONS:
Dietary Supplement: Hydrolyzed Collagen — Hydrolyzed collagen type II derived from the bone powder of Norwegian Atlantic salmon.
  Arms: Hydrolyzed Collagen type II
Other: Placebo — Pure maltodextrin.
  Arms: Maltodextrin
Dietary Supplement: CalGo — CalGo is a natural marine collagenic bone powder from salmon. The bone powder is a 100 % microcrystalline hydroxyapatite form of calcium and collagen type 2.
  Arms: Unhydrolyzed Collagen type II (Salmon bone meal)

SUMMARY:
The purpose of this study is to evaluate the efficacy of hydrolyzed collagen in osteoarthritis.

DETAILED DESCRIPTION:
The current study is part of a larger project called the CalGo-project. The overall purpose of the study is to use bone meal from salmon to promote skeletal health. Specifically, the potential for hydrolyzed collagen type II derived from salmon bone meal in ameliorating pain, stiffness and function in participants diagnosed with osteoarthritis will be evaluated over a time period of 6 months. Past literature indicates that collagen derivatives may be a potential supportive strategy in people suffering from osteoarthritis. Osteoarthritis is a common but complex joint disease with significant unmet medical needs, as there are currently no disease-modifying drugs available. Osteoarthritis represents a global health burden and the only curative treatment when pain becomes unmanageable, is joint replacement.

The dimensions of pain, stiffness, and function will be evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC 3.1). Plain x-rays with Kellgren-Lawrence grading will be employed to classify the severity of osteoarthritis. 100 potential participants will be screened for eligibility. Participants who meet the eligibility criteria will be randomized in a double-blind manner to receive 10 capsules daily of hydrolyzed collagen type II (a total of 5000 mg), 10 capsules daily of salmon bone meal, or 10 capsules daily of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Characteristic joint pain indicating osteoarthritis (OA) in the hip(s) or knee(s).
* A radiologically and clinically verified diagnosis of mild to moderate OA graded 1-3 on a Kellgren-Lawrence (KL) grading scale in affected hips or knees.
* Age 18-70 years.
* Familiar with the Norwegian language, both in writing and orally.
* Willingness to participate in the study.

Exclusion Criteria:

* A radiologically and clinically verified diagnosis of severe OA graded 4 on a KL grading scale in affected hips or knees.
* Use of drugs (and supplements) known to influence bone and joint metabolism, including Glucocorticoids, > 500 mg daily intake of elemental calcium in medication or supplement form, > 800 IU daily intake of vitamin D3, cancer therapy
* Pregnancy or breastfeeding
* Known fish allergy and history of hypersensitivity to any of the components in the interventional product.
* Other reasons which the principal investigator deems it necessary to exclude a potential participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline in WOMAC composite score at Month 3 and Month 6. | Baseline, 3 Months, and 6 Months
  A change in osteoarthritis symptomatology is assessed using a disease specific questionnaire (WOMAC 3.1).

SECONDARY OUTCOMES:
Mean change from from Baseline on the WOMAC pain subscale at Month 3 and Month 6. | Baseline, 3 Months, and 6 Months
  Pain is evaluated using the pain dimension of WOMAC 3.1, a disease-specific questionnaire. The pain subscale includes 5 items that assesses pain intensity. A score is produced when the value of each item is summarized. A higher score indicates worse pain.
Change from Baseline on an 11-point likert Global Assessment Scale at Month 3 and Month 6. | Baseline, 3 Months, and 6 Months
  A GAS scale gives an overall picture of an individuals' self-assessed effect of treatment. The individual is asked to compare the present health status with their health status at a previous point in time. The magnitude of this difference is scored numerically. In this study, we will use GAS on a 11-point Likert rating scale ranging from "completely recovered" to "worse than ever", with 0 being "unchanged" status.
Change from Baseline in pain intensity on a Numerical Rating Scale at Month 3 and Month 6. | Baseline, 3 Months, and 6 Months
  In this study, we will employ an 11-point (i.e., 0 to 10) Numerical Rating Scale as was recommended for use in chronic pain trials according to 2005 IMMPACT guidelines. 0 represents "No pain", and 10 represents "The most intense pain imaginable".
Change from Baseline in number of rescue medications self-administered during the study period. | Baseline, 6 Months
  Rescue medications that participants may use on an as needed basis include Paracetamol, typical NSAIDs, and analgesics containing opioids.
Change from Baseline in self-assessed quality of life on the EQ-5D-3L instrument at Month 3 and Month 6. | Baseline, 3 Months, and 6 Months
  EQ-5D-3L is a standardized instrument used to measure generic quality of life based on five distinct dimensions. EQ-5D-3L contains two parts. The first part contains five questions that the individual must answer and includes mobility (walking), self-care, usual activities, pain/discomfort, and anxiety/depression. For each item, there are three possible answers. Results are reported as a five-digit number ranging from 11111 (best health status) to 33333 (worst health status).
Difference in number of Adverse Events between the study groups. | 3 Months, and 6 Months.
  Reported between the hydrolyzed collagen group and placebo group, and the CalGo group and placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Bjerkestrand Lian, MD, PhD, Principal Investigator — Møre og Romsdal Hospital Trust (Helse Møre og Romsdal), Kristiansund Hospital
Locations (3):
- Norway (3):
  - Hofseth Biocare ASA, Ålesund, Møre og Romsdal
  - Kristiansund Hospital, Kristiansund, Møre og Romsdal
  - Lovisenberg Diakonale Sykehus, Oslo

IPD SHARING:
Plan to Share IPD: No